CLINICAL TRIAL: NCT01760902
Title: Diet & Activity Community Trial: High-Risk Inflammation
Acronym: CCTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, James hebert, James R. Hebert, MSPH, ScD, Director, University of South Carolina
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00001881; 5R24MD002769-02 (NIH)
Record Dates: First submitted 2012-12-12; First posted 2013-01-04 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Inflammation
Keywords: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diet and Physical Activity (Experimental): Participants convene weekly for 12 consecutive weeks and then once per month for 9 months. Each sessions is 90 minutes
  Interventions: Behavioral: Diet and Physical Activity

INTERVENTIONS:
Behavioral: Diet and Physical Activity — The group will convene weekly for 12 consecutive weeks and monthly thereafter for 9 consecutive months. Thus, there will be a total of 21 group-based sessions over the one-year period

SUMMARY:
South Carolina has many gaps in health status of our citizens. Some of the biggest gaps are higher cancer rates among African Americans. The purpose of this study is to find people who have increased inflammation and study how well a community-based dietary and physical activity program works at reducing the risk of African Americans developing inflammation-related diseases.

DETAILED DESCRIPTION:
A diet and physical activity intervention was developed to provide knowledge and skills to facilitate health behavior change in African-American Baptist Church members in South Carolina and promote healthy lifestyles to reduce colon cancer disparities. The intervention entitled, "H.E.A.L.S. (Healthy Eating and Active Living in the Spirit)" was used to train church education teams to deliver church and community educational activities promoting a diet rich in fruits and vegetables and an active lifestyle. The training focused leadership and empowerment skills to enable church lay leaders to become Church Education Teams (CETs) . The educational activities made it easier for church and community members to eat more fruits and vegetables, reduce fat intake, increase physical activity, and increase dietary intake of anti-inflammatory foods associated with colon cancer risk.

This 12 week healthy eating and physical activity program is tailored to meet a church's needs and goals by:

1. providing cooking classes, recipes,
2. tips for increasing the level of physical activity in their daily routine
3. assistance tracking basic measurements like

   * Weight
   * Blood pressure,
   * Inflammation levels

Education Goals:

* Increase knowledge of health behavior and changes that can impact health status
* Increase confidence in sharing health information with church, family, and community members.
* Develop skills to facilitate behavior change
* Develop skills to overcome barriers to behavior change

ELIGIBILITY:
Inclusion Criteria:

* African American

Exclusion Criteria:

* History of Cancer
* History of Ulcerative colitis
* Chrome Disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in C-Reactive Protein (CRP) levels from baseline to post intervention | Baseline, Post Intervention (90) days) and 12 months beyond baseline
  Data are collected at three time points: baseline, 90 days from baseline, and 12 months (one year) from baseline. Evaluable data will be difference from 90 days from baseline or 12 months (one year) from baseline or both.

SECONDARY OUTCOMES:
Change in Interleukin 6 (IL6) values from baseline to either 90 days or 12 months or both. | Baseline, Post intervention (90 days) and 12 months beyond baseline.
  As for the primary outcome measure, data are collected at three time points: baseline, 90 days from baseline, and 12 months (one year) from baseline. Evaluable data will be difference from 90 days from baseline or 12 months (one year) from baseline or both.
Change in body mass index (BMI) values from baseline to either 90 days or 12 months or both. | Baseline, Post intervention (90 days) and 12 months beyond baseline.
  As for the primary outcome measure, data are collected at three time points: baseline, 90 days from baseline, and 12 months (one year) from baseline. Evaluable data will be difference from 90 days from baseline or 12 months (one year) from baseline or both.
Change in body fat mass (BFM) values from baseline to either 90 days or 12 months or both. | Baseline, Post intervention (90 days) and 12 months beyond baseline.
  As for the primary outcome measure, data are collected at three time points: baseline, 90 days from baseline, and 12 months (one year) from baseline. Evaluable data will be difference from 90 days from baseline or 12 months (one year) from baseline or both.
Change in waist-to-hip ratio(WHR) values from baseline to either 90 days or 12 months or both. | Baseline, Post intervention (90 days) and 12 months beyond baseline.
  As for the primary outcome measure, data are collected at three time points: baseline, 90 days from baseline, and 12 months (one year) from baseline. Evaluable data will be difference from 90 days from baseline or 12 months (one year) from baseline or both.
Change in mcp-1 values from baseline to either 90 days or 12 months or both. | Baseline, Post intervention (90 days) and 12 months beyond baseline.
  As for the primary outcome measure, data are collected at three time points: baseline, 90 days from baseline, and 12 months (one year) from baseline. Evaluable data will be difference from 90 days from baseline or 12 months (one year) from baseline or both.

CONTACTS AND LOCATIONS:
Overall Officials: Jmaes R. Hebert, ScD, Principal Investigator — Universityof South Carolina
Locations (1):
- University of South Carolina (Columbia), Columbia, South Carolina, United States

REFERENCES:
- [Derived] Hebert JR, Wirth M, Davis L, Davis B, Harmon BE, Hurley TG, Drayton R, Angela Murphy E, Shivappa N, Wilcox S, Adams SA, Brandt HM, Blake CE, Armstead CA, Steck SE, Blair SN. C-reactive protein levels in African Americans: a diet and lifestyle randomized community trial. Am J Prev Med. 2013 Oct;45(4):430-40. doi: 10.1016/j.amepre.2013.05.011. PMID 24050419